CLINICAL TRIAL: NCT06766578
Title: Clinical Study of Low-dose Interval Radiotherapy Combined With Tirelizumab and SOX Chemotherapy Neoadjuvant Therapy for Locally Advanced Gastric/Gastroesophageal Junction Adenocarcinoma(STAR-02)
Brief Title: Clinical Study of Low-dose Interval Radiotherapy Combined With Tirelizumab and SOX Chemotherapy Neoadjuvant Therapy for Locally Advanced Gastric/Gastroesophageal Junction Adenocarcinoma
Acronym: STAR-02
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Li Leping, Professor, Shandong Provincial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NO.2024-1047
Record Dates: First submitted 2024-12-29; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Locally Advanced Gastric/Gastroesophageal Junction Adenocarcinoma
MeSH Terms: interventions — Oxaliplatin; S 1 (combination); Surgical Procedures, Operative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment arm(5×3Gy radiotherapy, tirelizumab, oxaliplatin, S-1) (Experimental)
  Interventions: Radiation: Neoadjuvant Therapy(5×3Gy radiotherapy); Drug: Neoadjuvant Therapy(tirelizumab, oxaliplatin, S-1); Procedure: Surgical treatment; Drug: Adjuvant therapy(SOX chemotherapy)

INTERVENTIONS:
Radiation: Neoadjuvant Therapy(5×3Gy radiotherapy) — Radiotherapy: 5×3Gy. The preoperative radiotherapy target was outlined by radiotherapy physicians according to the NCCN Guidelines for Gastric/esophagogastric Junction Tumor 2024 edition and the surgeon's opinions. The first and third cycles were 5×3Gy.
Drug: Neoadjuvant Therapy(tirelizumab, oxaliplatin, S-1) — The first and third cycles are 5×3Gy radiotherapy D1 to 5, intravenous administration for tirelizumab 200 mg D6, intravenous administration for oxaliplatin 130 mg/m2 D6, and oral administration twice a day for S-1 40 mg/m2 D6 to 19. The second and fourth cycles are intravenous administration for tirelizumab 200 mg D1, intravenous administration for oxaliplatin 130 mg/m2 D1, and oral administration twice a day for S-1 40 mg/m2 D1 to 14. Every treatment cycle is spaced 1 week apart.
Procedure: Surgical treatment — Surgical treatment is completed within 3-5 weeks after the end of neoadjuvant therapy.
Drug: Adjuvant therapy(SOX chemotherapy) — Postoperative adjuvant therapy is 4 cycles of SOX chemotherapy.

SUMMARY:
To evaluate the initial efficacy and safety of neoadjuvant low-dose interval radiotherapy combined with tirelizumab and SOX chemotherapy in locally advanced gastric/gastroesophageal junction adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients voluntarily participated in the study and signed informed consent with good compliance and follow-up;
* Adenocarcinoma of the gastric/gastroesophageal junction confirmed by endoscopic pathology (tumor located in the lesser bend of the stomach other than pylorus or the gastroesophageal junction) (Note: Pathology in other hospitals must be consulted by our hospital);
* Patients with cT4N+M0 AJCC stage 8 combined with endoscopic, CT, MRI, or PETCT findings;
* Age ≥18 years, ≤75 years, male and female;
* ECOG PS score 0-1;
* Presence of measurable and/or unmeasurable lesions as defined by the efficacy evaluation criteria for solid tumors (Recist 1.1);
* Has not received any prior systemic antitumor therapy (including but not limited to systemic chemotherapy, radiotherapy, molecular targeted drug therapy, immunotherapy, biotherapy, topical therapy, or other investigational therapeutic drugs;
* The functions of vital organs meet the following requirements (no blood components and cell growth factors are allowed to be used 2 weeks before screening) : Neutrophil absolute count (ANC) ≥ 1.5×10 9/L; Platelets ≥100×10 9/L; Hemoglobin ≥9g/dL; Serum albumin ≥2.8g/dL; Total bilirubin ≤ 1.5 ×ULN, ALT, AST and/or AKP≤2.5 ×ULN; serum creatinine ≤1.5 ×ULN or creatinine clearance ≥60mL/min (calculated according to the Cockcroft-Gault formula); International standardized ratio (INR) and activated partial thrombin time (APTT) ≤1.5×ULN (INR can be screened in the expected treatment range of anticoagulants for stable doses of anticoagulants such as low molecular weight heparin or warfarin);
* Fertile female subjects shall perform a urine or serum pregnancy test within 72 hours prior to receiving the first study drug, prove negative, and be willing to use an effective method of contraception during the trial period up to 5 months after the last drug administration.Male subjects whose partner is a woman of reproductive age should use an effective method of contraception during the trial period and for 7 months after the last dose.

Exclusion criteria

* a history of surgery for gastric/esophagogastric junction tumors;
* Previous history of fistula caused by primary tumor invasion;
* Higher risk of gastrointestinal bleeding and perforation;
* Poor nutritional status, BMI less than 18.5kg/m2, or PG-SGA score ≥9;
* Major surgery or severe trauma within 4 weeks prior to first use of the study drug;
* Uncontrolled pleural effusion, pericardial effusion or ascites requiring repeated drainage;
* has received or is currently receiving any of the following previous treatments: anti-PD-1 or anti-PD-L1 antibody therapy, chemotherapy, radiotherapy, targeted therapy;
* Received any investigational drug within 4 weeks prior to first use of the investigational drug;
* subjects requiring systemic treatment with corticosteroids (> 10mg prednisone equivalent daily dose) or other immunosuppressants within 2 weeks prior to initial use of the study drug, except for corticosteroids for esophageal/gastric local inflammation and for the prevention of allergy and nausea and vomiting.Other special circumstances, need to communicate with the bid. In the absence of active autoimmune disease, inhaled or topical steroids and adrenocorticosteroid replacement at doses > 10mg/ d of prednisone efficacy are permitted;
* those who have received antitumor vaccine or have received live vaccine within 4 weeks prior to the first administration of the study drug;
* have any active autoimmune disease or a history of autoimmune disease (such as interstitial pulmonary inflammation, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism); Except patients with vitiligo or recovered asthma/allergy of the same age without any intervention as adults;Patients with autoimmune mediated hypothyroidism treated with stable doses of thyroid hormone replacement and type 1 diabetes treated with stable doses of insulin could be included;
* have a history of immunodeficiency, including HIV positive, or other acquired or congenital immunodeficiency diseases, or have a history of organ transplantation or allogeneic bone marrow transplantation;
* any condition requiring systemic treatment with corticosteroids (more than 10 mg/ day of prednisone or its equivalent) or other immunosuppressant treatment within 14 days prior to treatment (except local, ocular, intraarticular, intranasal and inhaled corticosteroids with minimal systemic uptake); Prophylactic short-term (≤7 days) use of corticosteroids (e.g., to prevent contrast allergy) or for the treatment of non-autoimmune conditions (e.g., delayed hypersensitivity due to allergen exposure);
* subjects with uncontrolled cardiac clinical symptoms or disease, such as (1) NYHA II or above heart failure (2) unstable angina pecina (3) myocardial infarction within 1 year (4) clinically significant ventricular arrhythmias or ventricular arrhythmias requiring clinical intervention;
* Severe infection (CTCAE > level 2), such as severe pneumonia, bacteremia, and infectious complications requiring hospitalization, occurred within 4 weeks prior to initial use of the study drug; Chest imaging at baseline suggested active lung inflammation and signs and symptoms of infection requiring oral or intravenous antibiotic treatment within 2 weeks prior to enrollment, except for prophylactic antibiotic use;
* a history of interstitial lung disease, non-infectious pneumonia, pulmonary fibrosis or other uncontrolled acute lung disease;
* Patients with active pulmonary tuberculosis infection found by history or CT examination, or patients with active pulmonary tuberculosis infection history within 1 year before enrollment, or patients with active pulmonary tuberculosis infection history more than 1 year ago but without formal treatment;
* Subjects with active hepatitis B (HBV DNA≥2000 IU/mL or 10 4 Copies /mL), hepatitis C (positive hepatitis C antibody, and HCV-RNA higher than the lower limit of detection method);
* Abnormal values of sodium, potassium and calcium greater than grade 1 in laboratory tests within 2 weeks before enrollment, which could not be improved after treatment;
* known allergy to macromolecular protein preparations, or to any COMPONENT of PD-1, or allergy, hypersensitivity or contraindication to oxaliplatin or capecitabine or any component used in their preparations;
* A prior diagnosis of any other malignancy, other than malignancies with a low risk of metastasis and death (5-year survival > 90%), such as adequately treated basal or squamous cell skin cancer or carcinoma in situ of the cervix;
* pregnant or lactating women; Fertile subjects unwilling or unable to use effective contraception;
* According to the investigator's judgment, subjects have other factors that may cause them to be forced to terminate the study, such as other serious diseases (including mental diseases) requiring combined treatment, other recent serious diseases (such as myocardial infarction and cerebrovascular accident) with high risk of recurrence, seriously abnormal laboratory test values, family or social factors, which may affect subjects' safety or the collection of test data.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-12-31 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate (pCR) | From date of neoadjuvant therapy until the date of postoperative pathological assessment, assessed up to 16-18 weeks.
  Pathological complete response was defined as pT0N0M0

SECONDARY OUTCOMES:
Major pathological response rate (MPR) | From date of neoadjuvant therapy until the date of postoperative pathological assessment, assessed up to 16-18 weeks.
  The percentage of surviving tumor cells in the tumor bed after neoadjuvant therapy was ≤10%.
Objective response rate (ORR) | From date of neoadjuvant therapy until the date of surgery, assessed up to 15-17 weeks.
  Proportion of patients who achieved a complete response (CR) or a partial response (PR) as assessed by RECIST 1.1.
R0 resection rate | From date of neoadjuvant therapy until the date of postoperative pathological assessment, assessed up to 16-18 weeks.
  The proportion of patients who completed R0 resection in the total enrolled patients.
Treatment safety | From date of neoadjuvant therapy until the date of 30 days post-surgery, assessed up to 19-21 weeks.
  CTCAE 5.0 was used to record grade 3 and above treatment-related adverse reactions from the beginning of neoadjuvant therapy to 30 days after the end of surgery.
Postoperative complications | The first 30 days following surgery.
  Clavien-Dindo criteria were used to evaluate.
Event-free survival (EFS) | From date of neoadjuvant therapy until the date of the first occurrence of the above events, assessed up to 60 months.
  From the beginning of the study to the time of the first occurrence of any of the following events, disease progression beyond surgical treatment, local or distant recurrence, death from any cause, etc.
Overall survival (OS) | From the date of diagnosis to the date of death, assessed up to 60 months.
  From study inception to patient death from any cause.
Biomarkers | From the date of neoadjuvant therapy until the end of postoperative follow-up, assessed up to 60 months.
  By collecting tumor tissue and hematology samples before and after neoadjuvant therapy, scRNA-seq, WES, MRD and other techniques were used to explore biomarkers related to the efficacy of immunotherapy combined with radiotherapy and chemotherapy.

IPD SHARING:
Plan to Share IPD: Undecided